CLINICAL TRIAL: NCT00795730
Title: An Ascending Multiple Dose Study of the Safety, Pharmacokinetics, and Pharmacodynamics of NSA-789 Administered Orally to Healthy Subjects and Subjects With Alzheimer's Disease
Brief Title: Multiple Dose Study Evaluating the Safety and Tolerability of NSA-789
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wyeth is now a wholly owned subsidiary of Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3230A1-1002
Record Dates: First submitted 2008-11-20; First posted 2008-11-21 (Estimated); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Alzheimer Disease; Healthy Subjects
Keywords: Alzheimer's Disease; schizophrenia
MeSH Terms: conditions — Alzheimer Disease; Schizophrenia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Other: placebo
- NSA-789 (Experimental)
  Interventions: Drug: NSA-789

INTERVENTIONS:
Drug: NSA-789
  Arms: NSA-789
Other: placebo
  Arms: placebo

SUMMARY:
This is a multiple dose study of NSA-789, the purpose of which is to assess the safety and tolerability in healthy subjects and subjects with Alzheimer's Disease

ELIGIBILITY:
Inclusion Criteria

* Men or women aged 18 - 50 years (healthy subjects) or greater than 55 years old (subjects with Alzheimer's Disease)
* Women must be surgically sterile or postmenopausal
* Subjects with Alzheimer's Disease must be generally healthy, but may have a stable, chronic illness if well controlled.

Exclusion Criteria

* Healthy subjects may not be on any prescription or investigation drugs within 30 days of start of study.
* Subjects with Alzheimer's Disease may not be on any cholinesterase inhibitors such as donepezil (Aricept®) or rivastigmine (Exelon®) within 4 weeks of the start of the study.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Adverse event monitoring as specific tests that will be done to monitor safety (ECGs, certain laboratory tests, vital signs) and tolerability | 6 months

SECONDARY OUTCOMES:
Pharmacokinetic and pharmcodynamic parameters | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Wyeth is now a wholly owned subsidiary of Pfizer
Locations (1):
- Glendale, California, United States